CLINICAL TRIAL: NCT03814148
Title: Randomized, Double-blind, Double-dummy, National, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Leningrado 5 Association in the Treatment of Hypertension
Brief Title: Efficacy and Safety of Leningrado 5 Association in the Treatment of Hypertension
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The design of this protocol was rewritten due to regulatory recommendations.
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS0618-LENINGRADO 5
Record Dates: First submitted 2019-01-22; First posted 2019-01-23 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Arterial Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LENINGRADO 5 (Experimental): The study is double-dummy. Thus, the patient will take 2 tablets, as follow:
  1 tablet Leningrado 5 association and 1 tablet Natrilix® SR placebo.
  Interventions: Drug: LENINGRADO 5 association; Other: Natrilix SR Placebo
- Natrilix® SR (Active Comparator): The study is double-dummy. Thus, the patient will take 2 tablets, as follow:
  1 tablet Natrilix® SR 1,5 mg and 1 tablet Leningrado 5 association placebo.
  Interventions: Drug: Natrilix® SR; Other: Leningrado 5 association Placebo

INTERVENTIONS:
Drug: LENINGRADO 5 association — 1 coated sustained-release tablet, oral, once a day.
  Other Names: EMS association
  Arms: LENINGRADO 5
Drug: Natrilix® SR — 1 coated sustained-release tablet, oral, once a day.
  Other Names: Indapamide SR 1,5 mg
  Arms: Natrilix® SR
Other: Natrilix SR Placebo — 1 coated sustained-release tablet, oral, once a day.
  Other Names: Placebo
  Arms: LENINGRADO 5
Other: Leningrado 5 association Placebo — 1 coated sustained-release tablet, oral, once a day.
  Other Names: Placebo
  Arms: Natrilix® SR

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Leningrado 5 association on the treatment of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years or more;
* Participants diagnosed with hypertension, not controlled by monotherapy and/ or lifestyle modification;

Exclusion Criteria:

* Any clinical and laboratory findings that, in the judgment of the investigator, may interfere with the safety of research participants;
* BP ≥ 180/110 mmHg;
* Participants with BMI (body mass index) ≥ 40 Kg/m2;
* Previous diagnosis of secondary hypertension;
* History of Target Organ Injury;
* History of cardiovascular, hepatic and renal disease;
* History of gout, Diabetes Mellitus and hypokalemia;
* Current medical history of cancer;
* Current smoking;
* History of alcohol abuse or drug use;
* Pregnancy or risk of pregnancy and lactating patients;
* Known allergy or hypersensitivity to the medicines components used during the clinical trial;
* Participation in clinical trial in the year prior to this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Change in systolic blood pressure levels, as measured by ABPM at the initial visit and final visit. | 70 days

SECONDARY OUTCOMES:
Incidence and severity of adverse events recorded during the study | 101 days